CLINICAL TRIAL: NCT03506880
Title: Examining an Intervention to Reduce Underage DUI and Riding With Impaired Drivers
Brief Title: Project MADD - NIH Underage DUI and Ride
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Robert Turrisi, Professor of Biobehavioral Health, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 187458; R01AA025301 (NIH)
Record Dates: First submitted 2018-03-30; First posted 2018-04-24 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Underage Drinking; Driving Under the Influence; Drinking, Teen
MeSH Terms: conditions — Underage Drinking; Driving Under the Influence

STUDY DESIGN:
Intervention Model Description: 1 group receives the MADD parent intervention; the second group receives parent materials from the Surgeon General; and the third group is TAU
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MADD Materials (Experimental): Handbook developed by MADD and the PI to guide parents in discussing underage drinking, behaviors, and consequences with their teens
  Interventions: Behavioral: MADD Materials
- Surgeon General Materials (Experimental): Information published by the Surgeon General about teens and drinking
  Interventions: Behavioral: Surgeon General Materials
- Control (No Intervention): TAU

INTERVENTIONS:
Behavioral: MADD Materials — Handbook developed by MADD and the PI to guide parents in discussing underage drinking, behaviors, and consequences with their teens
  Arms: MADD Materials
Behavioral: Surgeon General Materials — Information published by the Surgeon General about teens and drinking
  Arms: Surgeon General Materials

SUMMARY:
Project MADD was designed to attempt to curb the alarming trends related to drunk driving and to move the field forward by testing a brief parent-intervention's ability to change adolescents' drinking, impaired driving, and riding with impaired driver behaviors. The aim of this project is to provide an easy-to-implement and low-cost alternative parent-based intervention that can be widely disseminated to address this important public health problem.

DETAILED DESCRIPTION:
Drunk driving is a major public health problem. The National Highway Traffic Safety Administration reported nearly 10,000 people died in alcohol-related crashes in the U.S. in 2014. The problem is further magnified when one considers that each year over 1.3 million drivers in the U.S. are arrested for alcohol-impaired driving. As alarming as these statistics are they pale by comparison to estimates indicating that they only represent 1% of the 121 million self-reported episodes of alcohol-impaired driving among U.S. drivers each year. The proposed research will attempt to curb these alarming trends and move the field forward by conducting a randomized controlled trial testing a brief parent intervention's ability to change adolescents' drinking, impaired driving, and riding with impaired driver behaviors. Prior brief parent-based interventions fro this lab have provided sufficient preliminary evidence of participation, communication, and efficacy for changing under-age drinking to warrant a large-scale comprehensive study. The study will use an extremely rigorous design that meets the Society for Prevention Research Criteria for Efficacy as described in Flay et al., a nationally representative sample assessed at 3-waves (baseline, 6 mo. and 12 mo.) to examine generalizability and sustained effects, and an oversampled Hispanic/Latino subgroup to examine the parent-intervention's potential to reduce a health disparity in an underserved population. The aims are as follows: Aim 1: Evaluate the efficacy of the parent intervention (short and long term); Aim 2: Examine mediators of the PBI that directly influence drinking, impaired driving, and riding with impaired driver behaviors; and Aim 3: Identify moderators to help inform future tailoring and improvement in intervention effectiveness. To the extent that the research is successful, it will provide an easy to implement and low cost alternative that can be widely disseminated to address this important public health problem.

ELIGIBILITY:
Inclusion Criteria:

* Parent and teen both consent (forming a dyad testing unit); They are part of GfK's KnowledgePanel pool of participants

Exclusion Criteria:

* Outside of the teen age range

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2352 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Turrisi, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parent-teen dyads were recruited from a nationally representative predetermined Web panel (KnowledgePanel, KP) maintained by the consumer company Ipsos. KP members were randomly selected through probability-based sampling of addresses from the U.S. Postal Services' Delivery Sequence File which covers approximately 97% of U.S. households. Only individuals who were sampled through these probability-based techniques were eligible to participate.
Groups:
- Active Control: Received HPV vaccine info
Period: Overall Study
Arm/Group | MADD Materials | Surgeon General Materials | Active Control
Started (The start of study enrollment included 1,176 parent-teen dyads. This means there were 1,176 enrolled in the study with 1,176 teens who completed the baseline survey.) | 393 | 393 | 390
T2 (30 -Days Post-baseline) (Only teen participants received the T2 baseline survey. 1,001 teen participants completed this survey.) | 331 | 328 | 342
T3 (6-months Post-baseline) (Parents and teens received the T3 survey. This means there were 952 parents and 952 teens who completed this survey.) | 315 | 318 | 319
T4 (12-months Post-baseline) (Parents and teens received the T4 survey. This means there were 906 parents and 906 teens who completed this survey.) | 296 | 305 | 305
Completed (The completed number reflects the number of parent-teen dyads who completed the study. There were 906 parents and 906 teens who completed this study.) | 296 | 305 | 305
Not Completed | 97 | 88 | 85

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MADD Materials | Surgeon General Materials | Active Control | Total
Number analyzed (Participants) | 393 | 393 | 390 | 1176
Age, Categorical [Count of Participants; unit: Participants]
  Teen Participants: <=18 years | 393 | 393 | 390 | 1176
  Teen Participants: Between 18 and 65 years | 0 | 0 | 0 | 0
  Teen Participants: >=65 years | 0 | 0 | 0 | 0
  Parent Participants: <=18 years | 0 | 0 | 0 | 0
  Parent Participants: Between 18 and 65 years | 385 | 387 | 382 | 1154
  Parent Participants: >=65 years | 8 | 6 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years]
  Teen Participants | 16.29 (1.09) | 16.37 (1.11) | 16.33 (1.09) | 16.33 (1.09)
  Parent Participants | 46.58 (7.44) | 46.90 (7.76) | 46.77 (7.65) | 46.75 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Teen Participants: Female | 179 | 197 | 203 | 579
  Teen Participants: Male | 214 | 196 | 187 | 597
  Parent Participants: Female | 223 | 213 | 204 | 640
  Parent Participants: Male | 170 | 180 | 186 | 536
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Teen Participants: Hispanic or Latino | 115 | 103 | 98 | 316
  Teen Participants: Not Hispanic or Latino | 278 | 290 | 292 | 860
  Teen Participants: Unknown or Not Reported | 0 | 0 | 0 | 0
  Parent Participants: Hispanic or Latino | 106 | 97 | 90 | 293
  Parent Participants: Not Hispanic or Latino | 287 | 296 | 300 | 883
  Parent Participants: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Teen Participants: American Indian or Alaska Native | 6 | 0 | 2 | 8
  Teen Participants: Asian | 15 | 12 | 13 | 40
  Teen Participants: Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Teen Participants: Black or African American | 32 | 35 | 33 | 100
  Teen Participants: White | 288 | 305 | 300 | 893
  Teen Participants: More than one race | 31 | 23 | 30 | 84
  Teen Participants: Unknown or Not Reported | 20 | 17 | 11 | 48
  Parent Participants: American Indian or Alaska Native | 5 | 2 | 7 | 14
  Parent Participants: Asian | 13 | 9 | 12 | 34
  Parent Participants: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Parent Participants: Black or African American | 32 | 31 | 39 | 102
  Parent Participants: White | 302 | 313 | 305 | 920
  Parent Participants: More than one race | 19 | 18 | 11 | 48
  Parent Participants: Unknown or Not Reported | 21 | 20 | 15 | 56
Teen Typical Weekly Drinking (DDQ) [Mean (Standard Deviation); unit: units on a scale] — Typical weekend drinking was assessed using the Daily Drinking Questionnaire (DDQ)[19], which asked teens to indicate the number of drinks they consumed on a typical Friday and Saturday during the past 6 months. These two items were summed to create the number of typical weekend drinks. Higher scores indicate the teen consumed a higher number of drinks on a typical weekend.
  units on a scale | 0.23 (0.97) | 0.20 (0.85) | 0.23 (1.01) | 0.22 (0.94)
Teen Riding with Impaired Drivers Measures [Mean (Standard Deviation); unit: units on a scale] — Impaired driving, declining to ride, and being a passenger in a car were assessed with 6 items (2 items for each sub-scale) adapted from Hultgren et al., 2018. Teens were asked to indicate the number of times they drove, declined a ride, or were a passenger with a drinking driver or driver who consumed drugs in the past 6 months. Responses were summed to indicate the number of times this occurred. Higher scores indicate the participant drove drunk (worse outcome), declined a ride (positive outcome), or were a passenger (worse outcome) more times.
  units on a scale
    Impaired driving | 0.16 (0.87) | 0.10 (0.68) | 0.08 (0.55) | 0.11 (0.71)
    Declining to ride with impaired driver | 0.51 (1.33) | 0.44 (1.32) | 0.37 (1.17) | 0.44 (1.28)
    Passenger in car with impaired driver | 0.57 (2.0) | 0.52 (1.82) | 0.46 (1.72) | 0.52 (1.85)

OUTCOME MEASURES:

1. Primary Outcome: Typical Weekend Drinking (DDQ)
Description: Typical weekend drinking was assessed using the Daily Drinking Questionnaire (DDQ; Collins et al., 1985), which asked teens to indicate the number of drinks they consumed on a typical Friday and Saturday during the past 6 months. These two items were summed to create the number of typical weekend drinks. Higher scores indicate the teen consumed a higher number of drinks on a typical weekend.
Time Frame: Baseline, 6 month follow-up, and 12 month follow-up
Population: Participants included in analyses from T4 (12-month post-baseline assessment).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MADD Materials | Surgeon General Materials | Active Control
Number analyzed (Participants) | 296 | 305 | 305
units on a scale | 0.53 (1.56) | 0.53 (1.57) | 0.38 (1.23)
Statistical Analysis 1: Comparison: MADD Materials vs Surgeon General Materials vs Active Control; It was hypothesized that drinking would increase from baseline to 12-month follow-up for those in the AC, but not for those in the SG and MADD conditions; Test type: Superiority; p > 0.05, Tukey's Post-Hoc; Mean Difference (Final Values) = 0.17 — Estimation parameter used to determine significance between mean values in MADD, SG, and AC group

2. Primary Outcome: Declining to Ride With Impaired Drivers
Description: Declining riding with impaired drivers was assessed with two items adapted from Hultgren et al (2018). Teens were asked to indicate the number of times they declined a ride from a driver that consumed alcohol and the number of times they declined a ride from a driver that consumed any drug other than alcohol (e.g., marijuana, opioids) in the past 6 months. Responses were summed to indicate the number of times they declined rides from impaired drivers in the past 6 months. Higher scores indicate the participant declined more rides from impaired drivers.
Time Frame: T4 (12-months post-baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MADD Materials | Surgeon General Materials | Active Control
Number analyzed (Participants) | 296 | 305 | 305
units on a scale | 0.61 (1.56) | 0.56 (1.38) | 0.31 (0.99)
Statistical Analysis 1: Comparison: MADD Materials vs Surgeon General Materials vs Active Control; It was also hypothesized that teens in the SG and MADD conditions would report significantly more declining rides with impaired drivers than those in the AC group; Test type: Superiority; p < 0.01, Tukey's Post-Hoc; Mean Difference (Final Values) = 0.16 — Estimation parameter used to determine significance between mean values in MADD, SG, and AC group

3. Secondary Outcome: Willingness to Ride in a Car With an Impaired Driver
Description: Willingness to ride in a car with an impaired driver was assessed with two items adapted from Hultgren et al. (2018). Teens responded using a 7-point scale that ranged from (0) Strongly disagree to (6) Strongly agree on their level of agreement to the following statements, "I am willing to be a passenger in a vehicle when the driver has consumed alcohol." and "I am willing to be a passenger in a vehicle when the driver has consumed any drug other than alcohol (e.g., marijuana, ecstasy, opioids).". Responses were averaged to create a mean score. Higher scores indicate the participant is more willing to be a passenger in a car with an impaired driver.
Time Frame: Baseline, 6 month follow-up, and 12 month follow-up
Population: Participants included in analyses from T3 (6-months post-baseline). These analyses examine participants willingness to ride in a car with an impaired driver.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MADD Materials | Surgeon General Materials | Active Control
Number analyzed (Participants) | 314 | 316 | 318
units on a scale | 1.22 (0.03) | 1.22 (0.03) | 1.22 (0.03)
Statistical Analysis 1: Comparison: MADD Materials vs Surgeon General Materials vs Active Control; It was hypothesized that participants in the MADD and SG groups would be significantly less willing to ride in a car with an impaired driver than those in the AC group; Test type: Superiority; p > 0.01, Tukey's Post-Hoc; Mean Difference (Final Values) = 0.06 — Estimation parameter used to determine significance between mean values in MADD, SG, and AC group

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | MADD Materials | Surgeon General Materials | Active Control
All-Cause Mortality (participants affected / at risk) | 0/393 | 0/393 | 0/390
Serious Adverse Events (participants affected / at risk) | 0/393 | 0/393 | 0/390
Other Adverse Events (participants affected / at risk) | 0/393 | 0/393 | 0/390

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT03506880/Prot_SAP_001.pdf